CLINICAL TRIAL: NCT00102791
Title: A Phase III Multicenter, 52-Week, Randomized, Double-Blind, Placebo-Controlled Study of the Clinical Efficacy and Safety of ICA-17043 With or Without HU Therapy in Patients With Sickle Cell Disease Who Have Had =>2 Acute Sickle-Related Painful Crises Within the Preceding 12 Months
Brief Title: A Stratified Sickle Event Randomized Trial (ASSERT)
Acronym: ASSERT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Because of the low probability of achieving the primary endpoint.
Sponsor: Icagen (Industry)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICA-17043-10
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2007-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — senicapoc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ICA-17043

SUMMARY:
The purpose of this study is to compare the effects of ICA-17043 to placebo with or without hydroxyurea (an oral drug used for treatment of sickle cell disease) in patients with sickle cell disease who have had 2 or more acute sickle-related painful crises requiring a visit to a medical facility within the past 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 65 years of age (inclusive)
* Male or female (not capable of becoming pregnant or using appropriate birth control)
* Medical history of sickle cell disease
* Have a history of at least two or more acute sickle-related painful crises requiring a visit to a medical facility within the preceding 12 months

Exclusion Criteria:

* Hemoglobin <4 or >11 g/dL
* On a chronic transfusion program
* Has significant active and poorly controlled (unstable) cardiovascular, neurologic, endocrine, hepatic, or renal disorders clearly unrelated to sickle cell disease

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2005-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Sickle Cell Crisis Rate | 52 weeks

SECONDARY OUTCOMES:
Time to First, Second, and Third Crisis | 52 Weeks
Maximum Crisis Morbidity Ranking | 52 Weeks
Efficacy Related Laboratory Parameters | 52 Weeks
Quality of Life | 52 Weeks
Health Economics | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Stocker, Ph.D., Study Director — Icagen
Locations (49):
- United States (42):
  - Mobile, Alabama
  - Little Rock, Arkansas
  - Davis, California
  - Los Angeles, California
  - Oakland, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Washington D.C., District of Columbia
  - Holly Hill, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Augusta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Brooklyn, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
- Brazil (3):
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Créteil, France
- Kingston, Jamaica
- Port of Spain, Trinidad and Tobago
- London, United Kingdom

REFERENCES:
- [Background] Stocker JW, De Franceschi L, McNaughton-Smith GA, Corrocher R, Beuzard Y, Brugnara C. ICA-17043, a novel Gardos channel blocker, prevents sickled red blood cell dehydration in vitro and in vivo in SAD mice. Blood. 2003 Mar 15;101(6):2412-8. doi: 10.1182/blood-2002-05-1433. Epub 2002 Nov 14. PMID 12433690
- See also: Icagen webpage — http://www.icagen.com